CLINICAL TRIAL: NCT03358017
Title: Multicenter, Randomized, Phase II Study of Neoadjuvant Chemotherapy Associated or Not With Zoledronate and Atorvastatin in Triple Negative Breast Cancers - YAPPETIZER Study
Brief Title: Neoadjuvant Zoledronate and Atorvastatin in Triple Negative Breast Cancer
Acronym: YAPPETIZER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mario Negri Institute for Pharmacological Research (Other)
Collaborators: Associazione Italiana per la Ricerca sul Cancro (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRFMN-BRC-7103; 2016-005112-17 (EudraCT Number)
Record Dates: First submitted 2017-11-13; First posted 2017-11-30 (Actual); Last update posted 2023-10-19 (Actual); Status verified 2023-10

CONDITIONS: Triple Negative Breast Cancer
Keywords: Triple negative breast cancer; Neoadjuvant chemotherapy; p53; Zoledronate; Atorvastatin; Mevalonate pathway inhibitors; Hippo pathway
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Zoledronic Acid; Atorvastatin

STUDY DESIGN:
Intervention Model Description: After providing informed consent for study participation, patients fulfilling the eligibility criteria will be randomized to receive standard anthracyclines/taxanes based neoadjuvant chemotherapy (ARM A) or the combination of zoledronate and atorvastatin associated with the above mentioned neoadjuvant chemotherapy (ARM B).
  Randomization will use a biased-coin minimization procedure having as stratification factor the type of neoadjuvant chemotherapy chosen by the center and the p53 level in the FFPE diagnostic core biopsy determined by IHC (<30% vs >30% vs unknown).
  Randomization and e-CFR will be handled by HeavyBase , an Open Source push based "peer to peer" electronic data management system.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARM A - standard NACT (Active Comparator): Standard anthracyclines/taxanes based neoadjuvant chemotherapy chosen by the investigator and administered according to clinical practice, for 6 months, or 4.5 months in case of dose dense schedule (unless disease progression, unacceptable toxicity, patient's refusal or investigator's decision)
  Interventions: Drug: Standard neoadjuvant cht
- ARM B - standard NACT + Zol + atorvastatin (Experimental): Standard anthracyclines/taxanes based neoadjuvant CT chosen by the investigator and administered according to clinical practice + Zoledronate 4 mg i.v. every 3-4 weeks and Atorvastatin 80 mg/die administered for 6 months, or 4.5 months in case of dose dense schedule (unless disease progression, unacceptable toxicity, patient's refusal or investigator's decision)
  Interventions: Drug: Zoledronate; Drug: Atorvastatin 80mg; Drug: Standard neoadjuvant cht

INTERVENTIONS:
Drug: Zoledronate — 4 mg i.v. every 3/4 weeks for 6 months
  Other Names: zoledronic acid
  Arms: ARM B - standard NACT + Zol + atorvastatin
Drug: Atorvastatin 80mg — 80mg /die os for 6 months
  Arms: ARM B - standard NACT + Zol + atorvastatin
Drug: Standard neoadjuvant cht — Standard neoadjuvant cht chosen by the investigator and administered according to clinical practice

SUMMARY:
Recent evidences suggest that zoledronate, one of the most used bisphosphonates (BPs) in the clinical setting for the prevention and treatment of bone metastasis in cancer patients, may have antitumor activity in early breast cancer. The ABCSG-12 clinical trial have reported improved Disease Free Survival (DFS) and Overall Survival (OS) in mostly chemotherapy naive premenopausal patients after a 3-years of treatment with zoledronate (zol) and ovarian-suppression therapy. The ZO-FAST study showed better DFS for immediate use of zol in postmenopausal patients receiving adjuvant hormonal treatment. Preliminary evidences support the role of zoledronate also in neoadjuvant setting reporting better responses in cases of treatment with zol and chemotherapy (cht) compared with cht alone. The anticancer mechanism of action of BPs still remains not well understood. Basically, BPs are mevalonate (MVA) pathway inhibitors and one of the most intriguing hypothesis supporting their anticancer activity relies on the modulation of the mevalonate downstream metabolism. Selected cancer subtypes may present a more pronounced mevalonate activity able to confer an aggressive phenotype. It has been shown that a mutant p53 acts as promoter of MVA upregulation. One of the most important biological implications of MVA pathway upregulation in cancer cells is the aberrant activation of the Hippo pathway, a molecular axis with a central role in carcinogenesis. Two Hippo pathway related transcriptional coactivators, YAP and TAZ, promote tissue proliferation and the self-renewal of normal and cancer stem cells, and incite metastasis. Due to the strong interplay between the MVA and Hippo pathways, the modulation of MVA axis has deep impact on the function of YAP/TAZ as transcriptional regulators of tumour growth. These findings implicate the mevalonate pathway as a therapeutic target for selected tumors with up-regulation of these pathways.

Preclinical and clinical evidences suggest that BPs are able to interfere with YAP/TAZ expression, via MVA pathway. This kind of activity may be part of the mechanism of action of BPs as antitumor drugs. Others medications are able to modulate the MVA pathway. Statins, a first-class of lipid-lowering medications that inhibit the enzyme HMG-CoA reductase, inhibit the sterol biosynthesis via the mevalonate pathway. A possible anti-tumor effect of statins can be predicted with the same mechanism of action described for BPs, through the interference with the MVA axis. Actually, the anti-tumor activity of statins have been investigated in different retrospective analyses. In breast cancer a more robust signal has been retrospectively reported and prospective studies have enquired the exquisite antitumor activity of statins in pre-operative breast cancer setting. From above, the clinical trial herein proposed aims to investigate the antitumoral clinical activity of zoledronate (zol) and statins (atorvastatin) combination, in patients receiving neoadjuvant chemotherapy for triple-negative breast cancer (TNBC). The primary objective of the study is to address in patients with TNBC the antitumor activity of pre-operative standard chemotherapy associated or not with zoledronate (zol) and atorvastatin measured through its effect on YAP and TAZ immunochemistry (IHC) expressions, which are considered co-primary objectives.

The primary clinical objective is to assess the anti-tumor activity of the combination of neoadjuvant standard cht associated with zol and atorvastatin, measured by the proportion of pCR obtained after neoadjuvant treatment in patients with TNBC.

Secondary objectives are: 1) to evaluate the anti-tumor activity of pre-operative standard chemotherapy associated or not with zol and atorvastatin according to high/low p53 levels 2) to address the efficacy of neoadjuvant cht associated or not with zol/atorvastatin combo in terms of disease free survival and overall survival); 3) to study the safety profile of study treatments; 4) to investigate the treatment modulation of YAP and TAZ gene expression (RNA-Seq) in tumor tissues collected at the time of core-biopsy and definitive surgery; 5) to address the modulation of Ki67expression by IHC in the FFPE diagnostic core biopsy tumor block and in the tumor tissue collected at surgery.

Patients fulfilling the eligibility criteria will be randomized to receive standard anthracyclines/taxanes based neoadjuvant cht (ARM A) or the combination of zol and atorvastatin associated with the above mentioned neoadjuvant cht (ARM B).

DETAILED DESCRIPTION:
Triple-negative breast cancer (TNBC) is a heterogeneous disease defined by the lack of expression of the estrogen receptor (ER), progesterone receptor (PR), and human epidermal growth factor receptor 2 (HER2). Roughly, it represents 15% of all breast cancers. Patients with TNBC are generally younger than the overall population of breast cancer patients and they are more frequently affected by larger and aggressive tumors (i.e. high nuclear-grading), associated with a poor prognosis and with a significant risk of relapse in the first three years after diagnosis. Since the negative expression of HER2 and hormone-receptors, patients affected by TNBC are not candidate for hormonal therapy or anti-HER2 agents, leaving cytotoxic chemotherapy as the only option for systemic therapy.

Despite these common features, TNBCs are characterized by a notable diversity within the group. Histologic variability provides one example of such diversity, with invasive ductal, metaplastic and medullary breast cancers (two very different subtypes of breast cancer) coexisting in this patient population. Furthermore, the TNBC subtype does not directly correspond to a single molecular breast cancer subgroup. Though most fit into the category of basal-like cancers, these groups are overlapping rather than synonymous, with certain populations of ER-positive and HER2-positive tumors also known to express basal-like markers. Indeed, molecular evaluation has identified additional subgroups within the TNBC, confirming the true heterogeneity and complexity of such subtype of breast cancer.

Due to this complex picture of histological and molecular characterization, TNBC still represents a therapeutic challenge for oncologist with several unmet clinical needs. Clearly, there is a need for a better understanding about the biology of TNBC and much more there is an urgent need for therapeutic options in TNBC, ideally in the form of targeted agents. Up to now, the heterogeneity of TNBC has made the achieving of these goals particularly complex. However, the identification of biomarkers able to predict response to systemic therapies is of crucial importance, as it will not only allow for better outcomes in responsive subgroups of TNBC, but also prevent unnecessary exposure of unresponsive patients to ineffective therapy. In this way, predictive biomarkers will facilitate the development of personalized medicine for TNBC.

At present, there is not a clear, proven effective single agent that targets a driving vulnerability in TNBC. However, there are a number of potential therapies currently under investigation that may eventually improve outcomes in these patients. Deep understanding of molecular pathways involved in TNBC carcinogenesis is of paramount importance for identify novel therapeutic options, including the optimal repositioning of drugs already available for clinical intent and potentially active in TNBC, such as the case of platinum salts, PARP-inhibitors (in BRCA mutation) and potentially bisphosphonates and statins, that represent the focus of this study.

Recent evidences suggest that zoledronate, one of the most used bisphosphonates (BPs) in the clinical setting for the prevention and treatment of bone metastasis in cancer patients, may have antitumor activity in early breast cancer. Clinical trials have shown some positive effects of BPs on patients outcome, reporting an improved Disease Free Survival (DFS) and Overall Survival (OS) in mostly premenopausal early breast cancer patients after a 3-years of treatment with zoledronate and ovarian suppression therapy and a better DFS for immediate use of zoledronate in postmenopausal patients receiving adjuvant hormonal treatment. Moreover, preliminary evidences support the role of zoledronate also in neoadjuvant setting with reported better responses in cases of treatment with zoledronate and chemotherapy compared with chemotherapy alone, suggesting a direct antitumor effect of zol in combination with cht.

In the final analysis of the AZURE trial no improvement in the primary endpoint of DFS was observed for the overall patient population. However, subgroup analysis showed that zoledronic acid significantly improved DSF (HR=0.76; p<0.005) in women who were at least 5 years postmenopausal at study entry. Moreover, zoledronate was found to improve overall survival including women of unknown menopausal status but with age older than 60 years.

In the same line of the neoAzure trial a more recently randomized clinical trial (the JONIE study) clearly confirmed the benefit of adding zol to neoadjuvant chemotherapy in HER2 negative early breast cancers. In that study Asian patients with HER2-negative invasive breast cancer were randomly assigned to either the CT or CT+ZOL (CTZ) group. One hundred and eighty-eight patients were randomized to either the CT group (n = 95) or the CTZ group (n = 93) from March 2010 to April 2012, and 180 patients were assessed. All patients received four cycles of FEC100 (fluorouracil 500 mg/m2, epirubicin 100 mg/m2, and cyclophosphamide 500 mg/m2), followed by 12 cycles of paclitaxel at 80 mg/m2 weekly. Zol (4 mg) was administered three to four times weekly for 7 weeks to the patients in the CTZ group. The primary endpoint was the pathological complete response (pCR) rate. The results of this randomized controlled trial indicated that the rates of pCR in CTZ group (14.8%) was doubled to CT group (7.7%), respectively (one-sided chi-square test, p = 0.068), though the additional efficacy of zoledronic acid was not demonstrated statistically. The pCR rate in postmenopausal patients was 18.4% and 5.1% in the CTZ and CT groups, respectively (one-sided Fisher's exact test, p = 0.071), and that in patients with triple-negative breast cancer was 35.3% and 11.8% in the CTZ and CT groups, respectively (one-sided Fisher's exact test, p = 0.112). The authors concluded the addition of zol to neoadjuvant CT has potential anticancer benefits in postmenopausal patients and in particular in the patients with triple-negative breast cancer. Actually, other clinical trials analyzed the role of BPs in breast cancer and, according to a recent meta-analysis of all randomized controlled trials (13 RCTs including more than 15.000 patients) that appraised the effects of BPs on survival irrespectively to the types of BPs, it seems evident a positive effect in selected patients (HR 0.81(0.69-0.95).

In line with this observation, Valachis A. et al. published a meta-analysis focusing on the specific role of zol as adjuvant treatment in breast cancer. In the meta-analysis fifteen studies were considered eligible and were further analyzed. The use of zol resulted in a statistically significant better overall survival outcome (five studies, 6,414 patients; hazard ratio [HR], 0.81; 95% confidence interval [CI], 0.70-0.94) while no significant differences were found for the disease-free survival outcome (seven studies, 7,541 patients; HR, 0.86; 95% CI, 0.70-1.06) or incidence of bone metastases (seven studies, 7,543 patients; odds ratio [OR], 0.94; 95% CI, 0.64-1.37).

Even though different explanations have been proposed over-time, the exact anticancer mechanism of action of BPs still remains not well understood. Basically, BPs are mevalonate (MVA) pathway inhibitors and one of the most intriguing hypothesis supporting their anticancer activity relies on the modulation of the mevalonate downstream metabolism. Mevalonate (MVA) is synthesized from 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) by HMG-CoA reductase (HMG-CoAR). MVA is further metabolized to farnesyl pyrophosphate (FPP), a precursor of cholesterol and sterols. FPP is also converted to geranylgeranyl pyrophosphate, and these lipids are used for post-translational modification of proteins that are involved in various aspects of tumor development and progression. Many studies showed that the MVA pathway is up-regulated in several cancers such as leukemia, lymphoma, multiple myeloma, as well as prostate, hepatic, pancreatic, esophageal and breast cancers. Several mechanisms may be involved in dysregulation of this pathway. They include mutation in HMG-CoAR and sterol-regulatory element binding protein (SREBP) and more specifically the mutation of p53. It has been shown that mevalonate pathway is significantly upregulated in case of mutant p53. Sterol biosynthesis intermediates reveal that this pathway is both necessary and sufficient for the phenotypic effects of mutant p53 on breast tissue architecture. It has been shown that the enzymes of the mevalonate pathways are under transcriptional control of SREBPs. In breast cancer cells oncogenic mutant p53 acts as a transcriptional cofactor for SREBPs, leading to elevated expression of mevalonate enzymes. One of the most important biological implications of MVA pathway upregulation in cancer cells is the aberrant activation of the Hippo pathway, a molecular axis with a central role in carcinogenesis. Two Hippo pathway related transcriptional coactivators, YAP and TAZ, promote tissue proliferation and the self-renewal of normal and cancer stem cells, and incite metastasis. Strikingly, YAP and TAZ are controlled by the same architectural features that first inhibit and then foster cancer growth, such as ECM elasticity, cell shape, and epithelial-to-mesenchymal transition. Due to the strong interplay between the MVA and the Hippo pathways, the modulation of MVA axis has deep impact on the function of YAP/TAZ as transcriptional regulators of tumour growth. These findings implicate the mevalonate pathway as a therapeutic target for selected tumors with up-regulation of these pathways.

Preclinical and clinical evidences, generated within the AIRC 5x1000 project, suggest that in selected breast cancer cases the BPs are able to interfere with YAP/TAZ expression, via MVA pathway. This kind of activity may be part of the mechanism of action of BPs as antitumor drugs.

Similarly to BPs, others medications are able to modulate the MVA pathway. Statins, also known as HMG-CoA reductase inhibitors, are a first-class of lipid-lowering medications that inhibit the enzyme HMG-CoA reductase, which plays a central role in the production of cholesterol. Statins inhibit the sterol biosynthesis via the mevalonate pathway. From above, a possible anti-tumor effect of statins can be predicted exactly with the same mechanism of action already described for BPs, i.e. through the interference with the MVA axis. Actually, the anti-tumor activity of statins have been investigated over-time in different retrospective analyses with conflicting results. In breast cancer a more robust signal has been retrospectively reported and, more recently, prospective studies have enquired the exquisite antitumor activity of statins in pre-operative breast cancer setting. Since BPs and statins act exactly on the same mevalonate pathway, a synergistic antitumor effect of the BPs and statins combination was predicted and reported in preclinical models, especially in cases of triple negative breast cancer, enriched in mutant p53 and YAP/TAZ expression.

From above, the clinical trial herein proposed aims to investigate the antitumoral clinical activity of zoledronate (zol) and statins (atorvastatin) combination, in patients receiving neoadjuvant chemotherapy for TNBC. The results of this project may eventually contribute to unveil a novel combined treatment in TNBC through the repositioning of clinical approved low toxic drugs, able to target relevant masterpieces of breast cancer cells metabolism.

The primary objective of the study is to address in patients with TNBC the antitumor activity of pre-operative standard chemotherapy associated or not with zoledronate (zol) and atorvastatin measured through its effect on YAP and TAZ immunochemistry (IHC) expressions, which are considered co-primary objectives (proof of concept objective).

The primary clinical objective is to assess the anti-tumor activity of the combination of neoadjuvant standard chemotherapy associated with zoledronate and atorvastatin, measured by the proportion of pathological complete response (pCR) obtained after neoadjuvant treatment in patients with TNBC.

Secondary objectives are: 1) to evaluate the anti-tumor activity of pre-operative standard chemotherapy associated or not with zoledronate (zol) and atorvastatin according to high/low p53 levels, measured through its effect on both YAP and TAZ IHC expressions and the proportion of pCR; 2) to address the efficacy of neoadjuvant chemotherapy associated or not with zoledronate/atorvastatin combo in terms of disease free survival (DFS) and overall survival (OS); 3) to study the safety profile of study treatments; 4) to investigate the treatment modulation (up/down regulation) of YAP and TAZ gene expression (RNA-Seq) in tumor tissues collected at the time of core-biopsy and definitive surgery; 5) to address the modulation of Ki67expression by IHC in the formalin fixed paraffin embedded (FFPE) diagnostic core biopsy tumor block and in the tumor tissue collected at surgery.

Patients fulfilling the eligibility criteria will be randomized to receive standard anthracyclines/taxanes based neoadjuvant chemotherapy (ARM A) or the combination of zoledronate and atorvastatin associated with the above mentioned neoadjuvant chemotherapy (ARM B).

The standard anthracyclines/taxanes based neoadjuvant CT will be administered according to the standard care in both arms; in the ARM B the neoadjuvant chemotherapy will be followed by zoledronate 4 mg i.v. (every 3/4 wks) and atorvastatin 80 mg/die, for a duration of 6 months of treatment (except for patients treated with dose- dense schedule who will receive zoledronate and atorvastatin for 4.5 months, according to the duration of neoadjuvant cht).

Prior to enrolment, the formalin fixed paraffin embedded (FFPE) diagnostic core biopsy specimens will be analyzed by investigational site pathologists to determine the presence of invasive TNBC and the p53 and Ki67 values by IHC. p53 and Ki67 evaluation will be then repeated at the time of definitive surgery. After enrolment, the FFPE diagnostic core biopsy will be tested for YAP and TAZ gene and protein expression by RNA-Seq and IHC respectively. The same evaluations will be then repeated at the time of definitive surgery.

The study is composed by two phases. Within the first phase patients will be randomized to one of the two study treatment arms described above. The relative reductions of YAP and TAZ IHC-expression at surgery with respect to core-biopsy analysis will be evaluated as primary proof of concept endpoint. The experimental arm containing zoledronate and atorvastatin will be considered deserving further development if a significant difference between arms in terms of relative reduction of YAP/TAZ IHC expression at surgery with respect to core-biopsy analysis will be identified in at least one of the two proteins. If such reduction in YAP or TAZ expression will be observed, at the second phase patients will be recruited only in the experimental arm (ARM B) and the control arm (ARM A) will be considered as calibration arm. Moreover the anti-tumor activity of the combination of neoadjuvant standard chemotherapy associated with zoledronate and atorvastatin measured by the proportion of patients with pCR obtained after neoadjuvant treatment will be assessed as primary clinical endpoint.

Patients will be monitored for AEs using the definitions and criteria for grading provided by NCI CTCAE version 4.03. Disease free survival (DFS) and overall survival (OS) will be assessed as secondary endpoints. The post treatment follow-up procedure required for all patients consists in disease assessment with mammography and breast ultrasound scan, according to RECIST criteria version 1.1, for the evaluation of the tumor burden and DFS, and visits following definitive surgery planned according to the clinical practice to report any new adverse events or changes in existing events in order to collect data on the secondary endpoints.

From 102 (1st phase) to 154 (2nd phase) patients will be registered in this clinical trial. The overall duration of the project, is expected to be 36 months, including 20 months for the execution of the first phase (recruitment, patients follow-up and data analysis), followed by 12 months for the running of the second phase. Fifteen experimental centers will take part into the study.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of non-metastatic operable TNBC subjected to diagnostic core biopsy
2. TNBC defined as HER2/ER/PgR negative receptors
3. Female, aged ≥ 18 years
4. ECOG (Eastern Cooperative Oncology Group) performance status ≤ 1
5. Clinical indication for a neoadjuvant approach according to the investigator's judgment. The standard chemotherapy will consist of a complete pre-operative treatment with anthracyclines and taxanes (in sequence or combination), including platinum derivatives and dose-dense schedules, according to the best physician choice (BPC)
6. Availability of paraffin-embedded tumor block (FFPE) taken at diagnostic biopsy for IHC and RNA-Seq molecular determinations
7. Patients with reproductive potential must have a negative serum pregnancy test within 7 days prior to study entry. They must agree to use a medically acceptable method of contraception throughout the treatment period and for 3 months after discontinuation of treatment
8. Written informed consent signed prior to enrolment according to ICH/GCP.

Exclusion Criteria:

1. Presence of metastatic disease
2. Previous investigational treatment for any condition within four weeks prior to study registration
3. Treatment with bisphosphonates, denosumab or other drug that, in the investigator's judgment, affects bone metabolism
4. Treatment with statins or other drugs that, in the investigator's judgment, potentially affect the mevalonate pathway
5. Any previous treatment for the currently diagnosed breast cancer, including radiation therapy, chemotherapy, biotherapy and/or hormonal therapy
6. Inadequate bone marrow, hepatic or renal function including the following:

   1. Hb< 9.0 g/dL, absolute neutrophil count < 1.5 x 109/L, platelets <100 x 109/L
   2. Total bilirubin > 1.5 x ULN, excluding cases where elevated bilirubin can be attributed to Gilberts Syndrome
   3. AST (SGOT), ALT (SGPT) > 2.5 x ULN
   4. Creatinine > 1.2 x ULN, calcium < 8.6 mg/dL
7. Co-existing active infection or concurrent illness that, at the judgment of the investigator, contra-indicate the inclusion of the patient in the study
8. Active liver disease or unexplained persistent elevations of serum transaminases exceeding 3 times the upper limit of normal
9. Co-existing dental diseases that form a contraindication to the use of zol
10. Any medical or other condition that in the Investigator's opinion renders the patient unsuitable for this study due to unacceptable risk
11. Psychiatric disorders or altered mental status precluding understanding of the informed consent process and/or completion of the necessary study assessment and procedures
12. Known hypersensitivity to the active substance, to other bisphosphonates or to any excipients of zoledronate
13. Known hypersensitivity to the active substance or to any excipients of atorvastatin. Conditions of rare hereditary problems of galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption
14. Anticipation of need for major surgical procedure during the course of the trial
15. Pregnant or breast feeding women.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 54 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2021-06-17 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
Proof of concept primary activity endpoint - Efficacy endpoint | At surgery, after 6 months of study treatment
  Relative reductions of YAP and TAZ IHC-expression at surgery with respect to core-biopsy analysis.
The proportion of responded patients | After 6 months of study treatment
  The clinical primary activity endpoint of the second phase of study is the proportion of responder patients, defined as those obtaining a pCR, defined as ypT0ypN0 or as the absence of any residual tumor burden at surgery.

SECONDARY OUTCOMES:
In relation to high/low p53 levels, relative reductions of YAP and TAZ IHC-expression at surgery with respect to core-biopsy analysis. Efficacy endpoint | At surgery, after 6 months of study treatment
  Relative reductions of YAP and TAZ IHC-expression at surgery with respect to core-biopsy analysis according to high/low p53 levels. A high level of p53 is defined by IHC expression ≥30%, while a low level by IHC expression <30%, as previously described
Proportion of responder patients according to high/low p53 levels - Efficacy endpoint | After 6 months of study treatment
  Proportion of responder patients according to high/low p53 levels
Disease Free Survival (DFS) - Efficacy endpoint | Date of first recurrence or relapse, second cancer, or death, whichever came first, assessed up to 36 months
  Disease free survival (DFS), defined as the time from the date of treatment start to the first of either recurrence or relapse, second cancer, or death, whichever comes first. Subjects alive not having relapse or recurrence or second cancer by the end of the study will be censored at the last disease assessment date.
Overall survival - Efficacy endpoint | Date of death from any cause, assessed up to 36 months
  Overall survival (OS), calculated for each patient as the time from the date of treatment start to the date of death from any cause. Patients not reported as having died at the end of the study will be censored at the date they were last known to be alive.
Regulation of YAP and TAZ gene expression by RNA-Seq in tumor tissue - Efficacy endpoint | At surgery, after 6 months of study treatment
  Proportions of patients with down regulation of YAP and TAZ gene expression by RNA-Seq in tumour tissue collected at definitive surgery with respect to tumour tissue collected at the time of core-biopsy for responder and non-responders patients.
Relative reduction of Ki67 in tumor samples - Efficacy endpoint | At surgery, after 6 months of study treatment
  Relative reduction of Ki67 IHC expression in tumour tissue samples collected at definitive surgery with respect to tumour tissue collected at the time of diagnostic core-biopsy for responder and non-responders patients.
Study treatment safety - Safety endpoint - AE | From the date of randomization/registration to the end of study, up to 36 months
  In order to address the safety endpoint the study will evaluate:
  - Incidence, nature, severity and seriousness of AEs, according of National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI CTCAE) version 4.03
Study treatment safety - Safety endpoint - Maximum grade | From the date of randomization/registration to the end of study, up to 36 months
  In order to address the safety endpoint the study will evaluate:
  - Maximum toxicity grade experienced by each patient for each specific toxicity
Study treatment safety - Safety endpoint - Percentage | From the date of randomization/registration to the end of study, up to 36 months
  In order to address the safety endpoint the study will evaluate:
  * Percentage of patients experiencing grade 3-4 toxicity for each specific toxicity
  * Percentage of patients with at least one SAE
  * Percentage of patients with at least one serious adverse drug reaction (SADR)
  * Percentage of patients with at least one suspect unexpected serious adverse reaction

CONTACTS AND LOCATIONS:
Overall Officials: Valter Torri, MD, Study Chair — Mario Negri Institute for Pharmacological Research Milano (Italy); Alberto Zambelli, MD, Principal Investigator — ASST Papa Giovanni XXIII, Bergamo, Italy
Locations (9):
- Italy (9):
  - Azienda Socio Sanitaria Territoriale ASST Lariana - Presidio Ospedaliero Ospedale S. Anna, San Fermo della Battaglia, Como
  - Azienda Socio Sanitaria Territoriale - ASST Papa Giovanni XXIII, Bergamo
  - Azienda Ospedaliero Universitaria di Bologna Policlinico S.Orsola - Malpighi, Bologna
  - Azienda Socio Sanitaria Territoriale - ASST di Cremona, Cremona
  - Azienda Socio Sanitaria Territoriale - ASST di Lodi, Lodi
  - Azienda Socio Sanitaria Territoriale Fatebenefratelli Sacco Sede Ospedale Fatebenefratelli, Milan
  - Azienda Socio Sanitaria Territoriale ASST Monza - Ospedale S. Gerardo, Monza
  - Istituti Clinici Scientifici Maugeri, Pavia
  - IFO - Istituto Nazionale dei Tumori Regina Elena, Roma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Foulkes WD, Smith IE, Reis-Filho JS. Triple-negative breast cancer. N Engl J Med. 2010 Nov 11;363(20):1938-48. doi: 10.1056/NEJMra1001389. PMID 21067385
- [Background] Reis-Filho JS, Tutt AN. Triple negative tumours: a critical review. Histopathology. 2008 Jan;52(1):108-18. doi: 10.1111/j.1365-2559.2007.02889.x. PMID 18171422
- [Background] Rakha EA, Elsheikh SE, Aleskandarany MA, Habashi HO, Green AR, Powe DG, El-Sayed ME, Benhasouna A, Brunet JS, Akslen LA, Evans AJ, Blamey R, Reis-Filho JS, Foulkes WD, Ellis IO. Triple-negative breast cancer: distinguishing between basal and nonbasal subtypes. Clin Cancer Res. 2009 Apr 1;15(7):2302-10. doi: 10.1158/1078-0432.CCR-08-2132. Epub 2009 Mar 24. PMID 19318481
- [Background] Lehmann BD, Bauer JA, Chen X, Sanders ME, Chakravarthy AB, Shyr Y, Pietenpol JA. Identification of human triple-negative breast cancer subtypes and preclinical models for selection of targeted therapies. J Clin Invest. 2011 Jul;121(7):2750-67. doi: 10.1172/JCI45014. PMID 21633166
- [Background] Oakman C, Viale G, Di Leo A. Management of triple negative breast cancer. Breast. 2010 Oct;19(5):312-21. doi: 10.1016/j.breast.2010.03.026. Epub 2010 Apr 10. PMID 20382530
- [Background] Gnant M, Mlineritsch B, Stoeger H, Luschin-Ebengreuth G, Heck D, Menzel C, Jakesz R, Seifert M, Hubalek M, Pristauz G, Bauernhofer T, Eidtmann H, Eiermann W, Steger G, Kwasny W, Dubsky P, Hochreiner G, Forsthuber EP, Fesl C, Greil R; Austrian Breast and Colorectal Cancer Study Group, Vienna, Austria. Adjuvant endocrine therapy plus zoledronic acid in premenopausal women with early-stage breast cancer: 62-month follow-up from the ABCSG-12 randomised trial. Lancet Oncol. 2011 Jul;12(7):631-41. doi: 10.1016/S1470-2045(11)70122-X. Epub 2011 Jun 5. PMID 21641868
- [Background] Bundred NJ, Campbell ID, Davidson N, DeBoer RH, Eidtmann H, Monnier A, Neven P, von Minckwitz G, Miller JC, Schenk NL, Coleman RE. Effective inhibition of aromatase inhibitor-associated bone loss by zoledronic acid in postmenopausal women with early breast cancer receiving adjuvant letrozole: ZO-FAST Study results. Cancer. 2008 Mar 1;112(5):1001-10. doi: 10.1002/cncr.23259. PMID 18205185
- [Background] Coleman RE, Winter MC, Cameron D, Bell R, Dodwell D, Keane MM, Gil M, Ritchie D, Passos-Coelho JL, Wheatley D, Burkinshaw R, Marshall SJ, Thorpe H; AZURE (BIG01/04) Investigators. The effects of adding zoledronic acid to neoadjuvant chemotherapy on tumour response: exploratory evidence for direct anti-tumour activity in breast cancer. Br J Cancer. 2010 Mar 30;102(7):1099-105. doi: 10.1038/sj.bjc.6605604. Epub 2010 Mar 16. PMID 20234364
- [Background] Coleman R, Cameron D, Dodwell D, Bell R, Wilson C, Rathbone E, Keane M, Gil M, Burkinshaw R, Grieve R, Barrett-Lee P, Ritchie D, Liversedge V, Hinsley S, Marshall H; AZURE investigators. Adjuvant zoledronic acid in patients with early breast cancer: final efficacy analysis of the AZURE (BIG 01/04) randomised open-label phase 3 trial. Lancet Oncol. 2014 Aug;15(9):997-1006. doi: 10.1016/S1470-2045(14)70302-X. Epub 2014 Jul 15. PMID 25035292
- [Background] Hasegawa Y, Tanino H, Horiguchi J, Miura D, Ishikawa T, Hayashi M, Takao S, Kim SJ, Yamagami K, Miyashita M, Konishi M, Shigeoka Y, Suzuki M, Taguchi T, Kubota T, Akazawa K, Kohno N; JONIE Study Group. Randomized Controlled Trial of Zoledronic Acid plus Chemotherapy versus Chemotherapy Alone as Neoadjuvant Treatment of HER2-Negative Primary Breast Cancer (JONIE Study). PLoS One. 2015 Dec 3;10(12):e0143643. doi: 10.1371/journal.pone.0143643. eCollection 2015. PMID 26633806
- [Background] Ben-Aharon I, Vidal L, Rizel S, Yerushalmi R, Shpilberg O, Sulkes A, Stemmer SM. Bisphosphonates in the adjuvant setting of breast cancer therapy--effect on survival: a systematic review and meta-analysis. PLoS One. 2013 Aug 26;8(8):e70044. doi: 10.1371/journal.pone.0070044. eCollection 2013. PMID 23990894
- [Background] Valachis A, Polyzos NP, Coleman RE, Gnant M, Eidtmann H, Brufsky AM, Aft R, Tevaarwerk AJ, Swenson K, Lind P, Mauri D. Adjuvant therapy with zoledronic acid in patients with breast cancer: a systematic review and meta-analysis. Oncologist. 2013;18(4):353-61. doi: 10.1634/theoncologist.2012-0261. Epub 2013 Feb 12. PMID 23404816
- [Background] Feldt M, Bjarnadottir O, Kimbung S, Jirstrom K, Bendahl PO, Veerla S, Grabau D, Hedenfalk I, Borgquist S. Statin-induced anti-proliferative effects via cyclin D1 and p27 in a window-of-opportunity breast cancer trial. J Transl Med. 2015 Apr 29;13:133. doi: 10.1186/s12967-015-0486-0. PMID 25925673
- [Background] Gobel A, Thiele S, Browne AJ, Rauner M, Zinna VM, Hofbauer LC, Rachner TD. Combined inhibition of the mevalonate pathway with statins and zoledronic acid potentiates their anti-tumor effects in human breast cancer cells. Cancer Lett. 2016 May 28;375(1):162-171. doi: 10.1016/j.canlet.2016.03.004. Epub 2016 Mar 8. PMID 26968247
- [Derived] Adams A, Jakob T, Huth A, Monsef I, Ernst M, Kopp M, Caro-Valenzuela J, Wockel A, Skoetz N. Bone-modifying agents for reducing bone loss in women with early and locally advanced breast cancer: a network meta-analysis. Cochrane Database Syst Rev. 2024 Jul 9;7(7):CD013451. doi: 10.1002/14651858.CD013451.pub2. PMID 38979716